CLINICAL TRIAL: NCT04130126
Title: Feasibility and Effects of Taking Cold Showers: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: eknz2019-00529
Record Dates: First submitted 2019-09-24; First posted 2019-10-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Sick Leave

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm showers (No Intervention): Participants in the warm showers condition are instructed to continue their normal warm showers throughout the study
- Cold showers (Experimental): Participants in the cold showers condition will be asked to take cold showers over a time period of 3 months
  Interventions: Behavioral: Taking cold showers

INTERVENTIONS:
Behavioral: Taking cold showers — Showering behaviour
  Arms: Cold showers

SUMMARY:
Considering the beneficial individual and environmental effects, investigators set out to replicate the recent study on the effects of taking cold showers on sickness absence, illness days and subjective well-being and to assess both the acceptability of taking cold showers as well as its effects on sickness absence and illness days as well as well-being, sleep quality, skin and hair appearance for a period of 3 months in a population of healthy and volunteering participants.

DETAILED DESCRIPTION:
The beneficial potential of cold-water immersion has been recognized throughout human history, with early references dating back to 1600 before Christ. These beneficial effects of the external application of cold water are also seen in more recent and more systematic approaches. Notably, cold water immersion had significant and positive effects on metabolic and catabolic processes, neurotransmitters and hormones, immune parameters as well as on more global markers of health, such as sick leave and quality of life. Also, cold showers have been proposed to be of use in the treatment of depression and there are anecdotal and uncontrolled reports as well as news coverage on taking cold showers - usually in contrast to warm or hot water - showing positive effects for skin and hair. For example, cold water tightens and constricts the blood flow which gives the skin and hair a healthier glow and decreases transepidermal water loss contributing to better skin hydration, while hot showers can lead to dried out skin. Noteworthy, none of these studies reported negative events related to cold water treatment as well as no negative long-term effects.

Furthermore, a recent study on 3018 healthy participants without any experience of cold showering and which were randomized to a (hot to-) cold shower for 30, 60, 90 seconds or normal (warm) showers for 30 days followed by 60 days of showering cold at their own discretion for the intervention groups - reported that 79% of participants taking cold showers completed the intervention protocol and that taking (hot to-) cold showers reduced sickness absence by 29% in comparison to participants taking normal hot showers (incident rate ratio: 0.71, P = 0.003). Importantly, no related serious adverse events were reported.

Next to these beneficial effects on health and well-being, taking cold showers has a rather neglected, but none the less important effect as taking cold showers substantially reduces individual CO2 emission. On the basis of the CO2 emission of the average electricity mix used in Switzerland (kwH=169g CO2) and the average habit of taking warm showers (Switzerland: 8.7 minutes 6 times per week, with 15 litres/minute of warm water of 35°C), taking warm water showers produces up to 248 kg of CO2 per person and year, which corresponds to a flight from Zurich to Paris and back. This CO2 emission per year significantly increases when the house-hold is run on natural gas (296 kg) or oil (390 kg). By ratifying the Paris Convention, Switzerland has committed itself to reducing greenhouse gas emissions by 50% by 2030 compared with 1990 levels. With the previously calculated example, 15% of per capita CO2 emissions could be saved to meet the 2030 target (25% if the house runs on oil; 19% on natural gas). Considering the urgent need to cut down CO2 emission, this neglected potential could be used to substantially reduce individual CO2 emission, besides achieving beneficial health and well-being effects.

Considering the beneficial individual and environmental effects, investigators set out to replicate the recent study on the effects of taking cold showers on sickness absence, illness days and subjective well-being and to assess both the acceptability of taking cold showers as well as its effects on sickness absence and illness days as well as well-being, sleep quality, skin and hair appearance for a period of 3 months in a population of healthy and volunteering participants.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants between 18 and 65 years of age
* no cold shower taken on a regular basis by participants

Exclusion Criteria:

* pregnant or lactating women
* subjects with cardiac, pulmonary or any other severe disease by self-report.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change of sickness absence | Assessed at baseline and then monthly for 3 months
  Sickness absence will be assessed at baseline and then monthly for 3 months. Participants are asked to retrospectively indicate the total number of days of absence from their work due to sickness. If participants indicate sickness absence over five days, they are asked for the reason.
Change in number of illness days | Assessed at baseline and then monthly for 3 months
  Illness days will be assessed at baseline and then monthly for 3 months. Participants are asked to retrospectively indicate the number of days that they have had symptoms of illness, cold or flu during the last month. If participants indicate illness over five days, they are asked for the reason.

SECONDARY OUTCOMES:
World Health Organization (WHO) Five Well-Being Index | Assessed at baseline and then monthly for 3 months
  The World Health Organization (WHO) Five Well-Being Index is a short questionnaire designed to measure well-being. The World Health Organization (WHO) Five Well-Being Index consists of five questions. The answers are given on a six-level scale (0 - 5, where 0 represents "No time at all" and 5 "All the time"). The raw value is obtained by adding the answers. The raw value ranges from 0 to 25, where 0 is the lowest quality of life and 25 is the highest quality of life. The percentage value of 0 -100 is obtained by multiplying by 4. The percentage value 0 denotes the worst state of health, 100 the best. The processing time is less than one minute. Example: In the last 4 weeks I was happy and in a good mood.
Questionnaire for positive aspects of well-being in adults | Assessed at baseline and then monthly for 3 months
  The Questionnaire for positive aspects of well-being in adults is a psychological self-evaluation procedure for the assessment of positive aspects of well-being in adults. The Questionnaire for positive aspects of well-being in adults consists of 16 questions, of which 4 questions each are assigned to one of the following four scales: Ability to work under pressure, vitality, enjoyment, inner peace. The answers are given on a 6-level scale (1 - 6, where 6 represents "Does not apply at all" and 1 "Is absolutely true"). The processing time is estimated at five to ten minutes by adding up the 16 items you get an overall result between 16 - 96, whereas a lower overall result shows a higher physical wellbeing. Example: There's hardly anything that can upset me.
International Physical Activity Questionnaire | Assessed at baseline and then monthly for 3 months
  The International Physical Activity Questionnaire is a short questionnaire designed to measure physical activity. The International Physical Activity Questionnaire consists of six questions, of which 3 questions each are assigned to one of the following two scales: Strong physical exertion and light physical exertion. Either you have to tick an answer or you will be asked for a time in hours and minutes per week. The processing time is estimated at three minutes. Example: If you are thinking about physical activities where you are at least a little out of breath, such as running, hiking, dancing, gardening or many sports, how many days a week do you do physical activities of this kind?
Pittsburgh Sleep Quality Index | Assessed at baseline and then monthly for 3 months
  The Pittsburgh Sleep Quality Index is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. The questionnaire offers seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is weighted on a 0-3 interval scale. The global Pittsburgh Sleep Quality Index score is then calculated by totalling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. Example: How tired are you during the day?
Skin quality questionnaire | Assessed at baseline and then monthly for 3 months
  The Skin quality questionnaire is a short self-report questionnaire that assesses hand and skin quality. The measure consists of 4 items, whereas they measure appearance, intactness, moisture con-tent and sensation on a 7-level scale, where higher scores denote a healthier quality of skin. The processing time is less than one minute each. Example: Appearance: Abnormal: redness, stains, rash. Normal: no redness, stains or rashes
Showering behaviour concerning frequency | Assessed at baseline and then weekly for 3 months
  At baseline, habitual showering behaviour will be assessed online and participants will rate their habitual showering behaviour in terms of frequency, duration, equipment (i.e. kind of shower head) and temperature. Participants are also asked to measure and indicate the temperature of their showers with a thermometer, but this is not obligatory for study continuation. After randomization, participants are asked to complete weekly online assessments of the showering behaviour for the duration of the study, i.e. frequency, duration, equipment (i.e. kind of shower head) and temperature. The intervention group is asked to shower for 3 months at the coldest level only, i.e. with water at the coldest level. The temperature of cold water will be estimated on the basis of average temperatures for the specific geographical region (which are obtained from local waterworks) and the dates of participation
Showering behaviour concerning duration | Assessed at baseline and then weekly for 3 months
  At baseline, habitual showering behaviour will be assessed online and participants will rate their habitual showering behaviour in terms of frequency, duration, equipment (i.e. kind of shower head) and temperature. Participants are also asked to measure and indicate the temperature of their showers with a thermometer, but this is not obligatory for study continuation. After randomization, participants are asked to complete weekly online assessments of the showering behaviour for the duration of the study, i.e. frequency, duration, equipment (i.e. kind of shower head) and temperature. The intervention group is asked to shower for 3 months at the coldest level only, i.e. with water at the coldest level. The temperature of cold water will be estimated on the basis of average temperatures for the specific geographical region (which are obtained from local waterworks) and the dates of participation
Showering behaviour concerning equipment | Assessed at baseline and then weekly for 3 months
  At baseline, habitual showering behaviour will be assessed online and participants will rate their habitual showering behaviour in terms of frequency, duration, equipment (i.e. kind of shower head) and temperature. Participants are also asked to measure and indicate the temperature of their showers with a thermometer, but this is not obligatory for study continuation. After randomization, participants are asked to complete weekly online assessments of the showering behaviour for the duration of the study, i.e. frequency, duration, equipment (i.e. kind of shower head) and temperature. The intervention group is asked to shower for 3 months at the coldest level only, i.e. with water at the coldest level. The temperature of cold water will be estimated on the basis of average temperatures for the specific geographical region (which are obtained from local waterworks) and the dates of participation
Showering behaviour concerning temperature | Assessed at baseline and then weekly for 3 months
  At baseline, habitual showering behaviour will be assessed online and participants will rate their habitual showering behaviour in terms of frequency, duration, equipment (i.e. kind of shower head) and temperature. Participants are also asked to measure and indicate the temperature of their showers with a thermometer, but this is not obligatory for study continuation. After randomization, participants are asked to complete weekly online assessments of the showering behaviour for the duration of the study, i.e. frequency, duration, equipment (i.e. kind of shower head) and temperature. The intervention group is asked to shower for 3 months at the coldest level only, i.e. with water at the coldest level. The temperature of cold water will be estimated on the basis of average temperatures for the specific geographical region (which are obtained from local waterworks) and the dates of participation

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gaab, Prof. Dr., Principal Investigator — Faculty for Psychology at the University of Basel
Locations (1):
- University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No